CLINICAL TRIAL: NCT01962272
Title: Randomised Trial of the Effects of Individual Nutritional Counseling in Cancer Patients
Brief Title: The Effect of Nutritional Counseling for Cancer Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Jens Rikardt Andersen, Associate Professor, Senior Physician, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-4-2009-135; H-4-2009-135 (Registry Identifier: Regional Ethics Commitee)
Record Dates: First submitted 2013-10-08; First posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Esophageal Cancer; Gastric Cancer; Uterine Cancer
Keywords: cancer; radiotherapy; chemotherapy; nutrition; dietary counseling; quality of life
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Uterine Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional counseling and Forticare® (Experimental): Weekly nutritional counseling and Forticare®. The goal being an intake that met the protein and energy requirements according to Harris-Benedict equation multiplied with an individual activity factor (1,1-1,5) and a stress factor (1,0-1,1). Daily protein requirements were estimated to 1,5 g/kg per day. In addition to the counseling, the patients in the intervention group were offered a high-protein nutrition supplement containing n-3 fatty acids (Forticare®, Nutricia). The recommended daily dose contained 2531 kJ, 33.8 g protein and 2.2 g EPA.
  Interventions: Behavioral: Weekly nutritional counseling; Dietary Supplement: Forticare®.
- Control (Active Comparator): The control group was nutritionally instructed by the nurses with the possibility to call for a dietician not related to the study if needed. No fixed schemes.
  Apart from the nutritional element the patients had the same care and therapy, including treatment of pain and side-effects to the treatment.
  Interventions: Behavioral: Weekly nutritional counseling

INTERVENTIONS:
Behavioral: Weekly nutritional counseling — The counseling included assessment of food intake, advice about improvement, motivation and specific food plans, as well as motivation to comply to the recommended dose of Forticare®.
Dietary Supplement: Forticare®.
  Arms: Nutritional counseling and Forticare®

SUMMARY:
Background and aims: Cancer-related malnutrition is multifactorial and related to a bad prognosis. The aim of this study was to investigate the effect of intensive, individual dietary counseling of patients in radiotherapy and/or chemotherapy for gynecologic-, gastric-, or esophageal cancer.

DETAILED DESCRIPTION:
The prospective, randomized controlled unblinded study with 61 consecutive outpatients. All patients were stratified according to primary disease (esophageal-, gastric- or gynecological cancer). Patients were randomised using tin foil-lined sealed envelopes by the authors. The sample size was calculated using 2α = 0.05, 1-β = 0.80, expected Standard Deviation (SD) (weight-loss-%) of 2.24 and the corresponding Minimal Relevant Difference of 1.75.

Due to different diagnoses and treatments, the duration of the participation in the study varied between 5 and 12 weeks (average 7.2 weeks). In all cases follow-up was performed three months after the end of treatment.

All patients randomized to receive nutritional intervention were counseled by the same dietitian at baseline, and once a week during treatment and at follow-up after three months. The goal of the nutritional counseling was an intake that met the protein and energy requirements according to Harris-Benedict equation multiplied with an individual activity factor (1,1-1,5) and a stress factor (1,0-1,1). Daily protein requirements were estimated to 1,5 g/kg per day. Dietary intake was evaluated by 24-hour-recall food questionnaires at baseline, every week, at the end of the study and at follow-up. On the basis of information from the 24-hour recall food questionnaires and supplementary comments patients were counseled on an individual basis with the purpose to minimize nutritional symptoms that may relate to cancer cachexia and the cancer treatment. The main elements of the counseling were to explain the importance of nutrition in relation to the patients present situation, to explain the targets and to agree on specific dietary goals to be fulfilled until the next session.

The control group was nutritionally instructed by the nurses with the possibility to call for a dietician if needed.

Apart from nutrition the patients had the same care and therapy, including treatment of pain and side-effects to the treatment.

The dietary data were coded and analysed for energy and protein content using a computerised version of Danish food composition tables.

In addition to the counseling, the patients in the intervention group were offered a high-protein nutrition supplement containing n-3 fatty acids (Forticare®, Nutricia). The recommended daily dose contained 2531 kiloJoule (kJ), 33.8 g protein and 2.2 g EPA. The use of dietary supplements and compliance with dietary recommendations were monitored weekly by questionnaire, interview and counting of residual containers with supplements. The data collection included recording of anthropometric data including body weight and body composition, biochemical nutritional status, nutritional status according to The Nutrition Risk Screening (NRS), and 24-hour dietary interview.

All participants were weighed at baseline, every week, at the end of the study and at follow-up. For a more detailed analysis of the weight development, Bioelectrical Impedance Analysis (BIA) was applied to assess the body composition of each patient. Measurements were performed by the investigators using an ElectroFluidGraph with a current (I) of 330 micro ampere (μA) and a frequency of 50 kilo herz (KHz) and according to Kyle and colleagues.

Quality of life (QoL) was measured at baseline, at the end of the study and at follow-up by using a self-administered questionnaire European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire QLQ-C30 version 3.0. This instrument is a 30- item cancer specific questionnaire designed to measure cancer patients' physical, psychological and social functions. This questionnaire was chosen because it has been shown to be reliable and valid in a number of studies. The questionnaire includes six function scales (physical, emotional, cognitive, social, role and global health), three symptom scales (fatigue, pain, nausea, or vomiting) and six single items assessing symptoms and the financial impact of the disease. A questionnaire developed in a previous study was used to assess treatment related side effects at the end of treatment by each patient. The questions covered the categories diarrhea, nausea, vomiting, loss of appetite, flatulence, abdominal pain and other kinds of pain.

The micronutrient status of the patients was assessed by blood analysis. The blood samples were obtained at baseline, at the end of treatment and at follow-up (p-Hemoglobin, p-Cobalamin, p-Ferritin, p-Transferrin, p-Iron, p-Magnesium, p-Phosphate, p-Albumin, p- Zinc).

ELIGIBILITY:
Inclusion Criteria:

* Adult, consecutive outpatients referred for either palliative or preoperative chemotherapy and/or radiation therapy of cancers in the stomach or the pelvic area.

Exclusion Criteria:

* Lack of ability to understand danish language and the instructions given

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Accumulated weight-change in per cent | up to 7.5 weeks
  The primary end-points were accumulated weight-loss or -gain in per cent of the weight measured between inclusion and end of treatment and between end of treatment and follow-up, respectively.

SECONDARY OUTCOMES:
Treatment related side effects and Quality of Life | up to 7.5 weeks
  Secondary endpoints were treatment related side effects and Quality of Life.

CONTACTS AND LOCATIONS:
Overall Officials: Jens R Andersen, MD,MPA, Principal Investigator — University of Copenhagen
Locations (1):
- Departmen of Oncology, Rigshospital, Copenhagen, Denmark